CLINICAL TRIAL: NCT06704542
Title: A Study of the Impact of Abnormal Glucose Tolerance in Allogeneic Hematopoietic Stem Cell Transplantation Donors on Recipients' Post-Transplant Survival Outcomes: A Multicenter Retrospective Cohort Study Based on HIS Data
Brief Title: Abnormal Glucose Tolerance in Allogeneic Hematopoietic Stem Cell Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Xiaoxia, Director of the Center for Translational Medicine, Ruijin Hospital
Other Study IDs: RJBMT-07
Record Dates: First submitted 2024-11-13; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION; Diabetes Mellitus; Impaired Fasting Glucose
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 1. Peripheral blood/bone marrow specimens from post-transplant patients. 2. Peripheral blood stem cell grafts from donors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: patients who underwent allogeneic hematopoietic stem cell transplantation from March 2019 to March 2024; donor fasting blood glucose and/or HbA1c data available; fasting blood glucose ≥6.1 mmol/L or HbA1c ≥5.7%
- Control Group: patients who underwent allogeneic hematopoietic stem cell transplantation from March 2019 to March 2024; donor fasting blood glucose and/or HbA1c data available; fasting blood glucose <6.1 mmol/L; HbA1c <5.7% (if available)

SUMMARY:
To investigate the impact of abnormal glucose tolerance in hematopoietic stem cell transplantation donors on patients' post-transplant survival outcomes.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is an important means of treating a variety of hematologic disorders. With the progress of HSCT technology, especially the research on haploidentical transplantation (HID-HSCT), the range of donor choices for hematological patients has been expanded, and theoretically, the era of "everyone has a donor" has been reached, which has increased the chances for hematological patients to receive allo-HSCT . The efficacy of allo-HSCT has improved dramatically over the past decades, but post-transplant complications such as graft-versus-host disease (GvHD), infections, and disease recurrence may still lead to treatment failure. In order to improve the efficacy of allo-HSCT, in addition to the improvement of pretreatment regimen and post-transplant management, the selection of the best donor among the many alternatives (including sibling donors, parents, children, and collateral hematologic donors, etc.) is still the focus and difficulty of clinical decision-making. The existing studies on donor selection have suggested that the factors to be considered include the number of HLA mismatched sites, donor-recipient consanguinity, donor age and gender, donor-specific antibody (DSA), NK cell isotype reactivity, and clonal hematopoiesis of the donor . However, little is known about whether a donor with metabolic syndrome such as diabetes affects post-transplant survival in allo-HSCT recipients.

It has been shown that diabetes mellitus affects the number and function of hematopoietic and immune cells, and that these effects may be passed on to progeny blood cells through epigenetic mechanisms, with long-term effects on immune cell function in diabetic patients. We therefore hypothesized that the effects of abnormal glucose metabolism in donors on the hematopoietic system may affect hematopoiesis and immune reconstitution in transplant recipients through "metabolic memory". Therefore, the investigator conduct a multicenter retrospective study through multifactorial survival regression. It is expected to provide new theoretical support for optimizing donor selection for allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent allogeneic hematopoietic stem cell transplantation (HSCT) between March 2019 and March 2024;
* Donor had fasting blood glucose and/or HbA1c records
* Eastern Cooperative Oncology Group (ECOG) physical fitness score of 0-2
* Survived at least 12 weeks after HSCT
* Voluntarily signed the Informed Consent Form
* Had appropriate organ function;
* Laboratory results within 7 days prior to HSCT met the following criteria:

  1. Aspartate aminotransferase (AST) ≤ 3-fold (upper limit of norma, ULN);
  2. Alanine aminotransferase (ALT) ≤ 3x ULN;
  3. Total serum bilirubin ≤ 1.5 times the upper limit of normal ULN unless the patient has documented Gilbert syndrome; patients with Gilbert-Meulengracht syndrome with bilirubin ≤ 3.0 times the upper limit of normal and direct bilirubin ≤ 1.5 times the upper limit of normal may be included;
  4. Serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 60 mL/min;
  5. Coagulation function: International Normalized Ratio (INR) ≤1.5×ULN, Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN;

Exclusion Criteria:

* Active autoimmune diseases such as SLE, rheumatoid arthritis, etc.
* Active cardiovascular disease such as uncontrolled arrhythmias, uncontrolled hypertension, congestive heart failure, any Grade 3 or 4 heart disease as determined by the New York Heart Association (NYHA) Functional Class, or a history of myocardial infarction in the 6 months prior to screening;
* Other serious medical conditions that may limit the patient's participation in this trial (e.g., progressive infection, uncontrolled diabetes);
* HIV infection, or chronic infection with hepatitis B virus (HBsAg-positive) or hepatitis C virus (anti-HCV-positive) that cannot be controlled by medications;
* Patients with other uncured tumors
* Patients with neurological or psychiatric disorders
* Patients who were unable to understand or comply with the research protocol or are unable to sign the Informed Consent Form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were diagnosed with hematological disorders and underwent allo-HSCT
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | One year-overall survival since hematopoietic stem cell transplantation
  Patient's overall survival time since hematopoietic stem cell transplantation

SECONDARY OUTCOMES:
Non-relapse Mortality (NRM) | One year since hematopoietic stem cell transplantation
  NRM after hematopoietic stem cell transplantation
Relapse-free Survival (RFS) | One year since hematopoietic stem cell transplantation
  RFS after hematopoietic stem cell transplantation
Event-free Survival (EFS) | One year since hematopoietic stem cell transplantation
  EFS after hematopoietic stem cell transplantation
Graft versus Host Disease (GvHD) incidence | One year since hematopoietic stem cell transplantation
  GvHD incidence after hematopoietic stem cell transplantation
GvHD and Relapse-free Survival (GRFS) | One year since hematopoietic stem cell transplantation
  GRFS incidence after hematopoietic stem cell transplantation
Cumulative Incidence Rate (CIR) | One year since hematopoietic stem cell transplantation
  CIR after hematopoietic stem cell transplantation
Graft Time of Different Cell Subpopulation | One year since hematopoietic stem cell transplantation
  Graft Time of Platelet, Neutrophil

CONTACTS AND LOCATIONS:
Overall Officials: Jingtao Huang, Principal Investigator — Ruijin Hospital
Locations (6):
- China (6):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital of Huazhong University of Science and Technology, Wuhan, Wuhan, Hubei
  - Li Quan Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - The First Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Hospital of Hematology of the Chinese Academy of Medical Sciences, Tianjin

IPD SHARING:
Plan to Share IPD: No